CLINICAL TRIAL: NCT03295357
Title: Extubation of Patients on ECLS is Associated With a Reduction in Complications Related to Mechanical Ventilation: Retrospective Single-centre Study
Acronym: EXTUB ECLS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: LAMIREL-GIRARD 2016
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Extra-Corporeal Life Support

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with extubation while on ECLS
- Patients without extubation

SUMMARY:
There are no clear recommendations concerning the management of patients on ECLS (Extra-Corporeal Life Support). Many teams keep patients sedated until removal of the ECLS so as to avoid accidents, notably decannulation. Moreover, there are few publications on the subject, all the more so as the extubation of patients on ECLS (Extra-Corporeal Life Support) is a recent practice. Nonetheless, it is becoming more and more frequent in the cardiovascular ICU of Dijon University Hospital. We therefore wished to evaluate the benefits of this practice by comparing 2 populations: those with extubation while on ECLS (Extra-Corporeal Life Support) and those without.

ELIGIBILITY:
Inclusion Criteria:

- Patients over 18 years who were placed on ECLS between 1/01/14 and 31/12/15

Exclusion Criteria:

* Patients under 18 years old
* Patients on ECLS for a heart transplant
* Patients who died within the first 48 hours following the initiation of ECLS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on ECLS
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of VAP (ventilator-associated pneumonia) during hospitalisation in the ICU | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France